CLINICAL TRIAL: NCT04491552
Title: TruGraf® Long-term Clinical Outcomes Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TGRP06
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Kidney Transplant Rejection
Keywords: Biomarkers; Subclinical Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients monitored with TruGraf and TRAC testing: Subjects will have TruGraf and TRAC testing at study enrollment (Baseline) and thereafter every 3 months. In addition subjects will have TRAC testing at any time there is a suspicion of acute rejection.
  Interventions: Diagnostic Test: Patients monitored with TruGraf and TRAC testing

INTERVENTIONS:
Diagnostic Test: Patients monitored with TruGraf and TRAC testing — This is an observational study there are no protocol mandated interventions. TruGraf and TRAC results will be utilized in conjunction with standard of care assessments to determine patient management.

SUMMARY:
This is a prospective, multi-center, observational study. Subjects will have OmniGraf™ (TruGraf® and TRAC™) testing at study enrollment and thereafter every 3 months. In addition subjects will have OmniGraf™ (TruGraf® and TRAC™) testing at any time there is a clinical suspicion of acute rejection. Data collection for the primary objective extends over a 2-year period.

DETAILED DESCRIPTION:
Several studies have validated TruGraf® in stable renal transplant patients to rule out subclinical acute rejection. These studies generally evaluated the diagnostic value of TruGraf® at single timepoints. Thus the value of serial monitoring and changes over time has not been previously investigated. In addition, no study has assessed TruGraf® and TRAC™in a serial and longitudinal fashion.

Therefore the aim of this study is to evaluate the impact of serial monitoring renal transplant patients with both TruGraf® and TRAC™ on long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization;
* At least 18 years of age;
* Recipient of a primary or subsequent deceased-donor or living-donor kidney transplant;
* At least 3-months post-transplant;
* Stable serum creatinine (per Principal Investigator);
* Treated with any immunosuppressive regimen, and;
* Selected by provider to undergo OmniGraf™ (TruGraf® and TRAC™) testing as part of post-transplant care; and

Exclusion Criteria:

* Recipient of a combined organ transplant with an extra-renal organ and/or islet cell transplant;
* Recipient of a previous non-renal solid organ and/or islet cell transplant;
* Known to be pregnant;
* Known to be infected with HIV;
* Known to have Active BK nephropathy;
* Known to have nephrotic proteinuria (Per Principal Investigator);
* Participation in other biomarker studies testing clinical utility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an observational study in adult (age ≥ 18 years), kidney transplant patients who are at least one year from the time of transplant. Approximately 2000 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
occurrence of either biopsy proven acute rejection (BPAR) on a for cause biopsy or graft loss, or a decrease from baseline in eGFR > 10 mL/min. | Baseline to month 24

SECONDARY OUTCOMES:
First occurrence of biopsy proven acute rejection (on a for cause biopsy) | Baseline to month 24
First occurrence of clinically treated acute rejection | Baseline to month 24
Proteinuria | Baseline to month 24
  defined by a spot urine protein-creatinine ratio > 0.5
TruGraf results | Baseline to month 24
  The proportion of TruGraf not-TX results
TRAC results | Baseline to month 24
  The proportion of TRAC results > 0.69
Clinical Utility of TruGraf and TRAC in clinical decision making | Baseline to month 24
  Percent of total number of TruGraf results that the PI identified as having clinical utility
Proportion of subjects who develop de novo donor-specific HLA antibodies class I and class II (dnDSA) | Baseline to month 24
  Proportion of subjects who develop de novo donor-specific HLA antibodies class I and class II (dnDSA)
Proportion of subjects with graft loss | Baseline to month 24
  defined as permanent return to dialysis, retransplantation or patient death at any time during the 2-year primary follow-up study period
Graft survival | Baseline to month 24
  calculated from the date of kidney transplantation until data of graft loss
Proportion of subjects with death-censored graft loss | Baseline to month 24
  defined as permanent return to dialysis or retransplantation at any time during the 2-year primary follow-up study period. Patients who die with a functioning graft will be right censored
Percent subject death period | Baseline to month 24
  Subject death from any cause at any time
Subject survival | Baseline to month 24
  calculated from date of kidney transplantation until date of patient death
Estimated GFR | Baseline to month 24
  calculated using the MDRD 4-variable equation

CONTACTS AND LOCATIONS:
Overall Officials: Patty W. Thielke, PharmD, Principal Investigator — Transplant Genomics, Inc.
Locations (36):
- United States (36):
  - Banner University Medical Center Tucson, Tucson, Arizona
  - Fresno Nephrology Medical Group, Fresno, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - House of Transplant and Cancer- Riverside Community Hospital, Riverside, California
  - University of California Davis, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Illinois-Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - Universtiy of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Renal and Transplant Associates of New England, Springfield, Massachusetts
  - Primary Coordinator Coordinator, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Erie County Medical Center, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - UR Medicine Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Clinical Research Strategies, Houston, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Primary Coordinator, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Boyle G, Snyder JJ, Kasiske BL, Israni AK. Kidney. Am J Transplant. 2016 Jan;16 Suppl 2(Suppl 2):11-46. doi: 10.1111/ajt.13666. PMID 26755262
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Rush D, Nickerson P, Gough J, McKenna R, Grimm P, Cheang M, Trpkov K, Solez K, Jeffery J. Beneficial effects of treatment of early subclinical rejection: a randomized study. J Am Soc Nephrol. 1998 Nov;9(11):2129-34. doi: 10.1681/ASN.V9112129. PMID 9808101
- [Background] El Ters M, Grande JP, Keddis MT, Rodrigo E, Chopra B, Dean PG, Stegall MD, Cosio FG. Kidney allograft survival after acute rejection, the value of follow-up biopsies. Am J Transplant. 2013 Sep;13(9):2334-41. doi: 10.1111/ajt.12370. Epub 2013 Jul 19. PMID 23865852
- [Background] Loupy A, Vernerey D, Tinel C, Aubert O, Duong van Huyen JP, Rabant M, Verine J, Nochy D, Empana JP, Martinez F, Glotz D, Jouven X, Legendre C, Lefaucheur C. Subclinical Rejection Phenotypes at 1 Year Post-Transplant and Outcome of Kidney Allografts. J Am Soc Nephrol. 2015 Jul;26(7):1721-31. doi: 10.1681/ASN.2014040399. Epub 2015 Jan 2. PMID 25556173
- [Background] First MR, Pierry, D, McNultuy, M et al. Analytical and clinical validation of a molecular diagnostic signature in kidney transplant recipients. J Transplant. Technol. Res. 2017; 7(3).
- [Background] US Renal Data System. 2016 USRDS annual data report: Epidemiology of kidney disease in the United States. Bethesda, MD: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2016.
- [Background] Marsh CL, Kurian SM, Rice JC, Whisenant TC, David J, Rose S, Schieve C, Lee D, Case J, Barrick B, Peddi VR, Mannon RB, Knight R, Maluf D, Mandelbrot D, Patel A, Friedewald JJ, Abecassis MM, First MR. Application of TruGraf v1: A Novel Molecular Biomarker for Managing Kidney Transplant Recipients With Stable Renal Function. Transplant Proc. 2019 Apr;51(3):722-728. doi: 10.1016/j.transproceed.2019.01.054. Epub 2019 Jan 26. PMID 30979456
- [Background] Snyder TM, Khush KK, Valantine HA, Quake SR. Universal noninvasive detection of solid organ transplant rejection. Proc Natl Acad Sci U S A. 2011 Apr 12;108(15):6229-34. doi: 10.1073/pnas.1013924108. Epub 2011 Mar 28. PMID 21444804
- [Background] De Vlaminck I, Martin L, Kertesz M, Patel K, Kowarsky M, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Nicolls MR, Cornfield D, Weill D, Valantine H, Khush KK, Quake SR. Noninvasive monitoring of infection and rejection after lung transplantation. Proc Natl Acad Sci U S A. 2015 Oct 27;112(43):13336-41. doi: 10.1073/pnas.1517494112. Epub 2015 Oct 12. PMID 26460048
- [Background] Gielis EM, Ledeganck KJ, De Winter BY, Del Favero J, Bosmans JL, Claas FH, Abramowicz D, Eikmans M. Cell-Free DNA: An Upcoming Biomarker in Transplantation. Am J Transplant. 2015 Oct;15(10):2541-51. doi: 10.1111/ajt.13387. Epub 2015 Jul 16. PMID 26184824
- [Background] Sharon E, Shi H, Kharbanda S, Koh W, Martin LR, Khush KK, Valantine H, Pritchard JK, De Vlaminck I. Quantification of transplant-derived circulating cell-free DNA in absence of a donor genotype. PLoS Comput Biol. 2017 Aug 3;13(8):e1005629. doi: 10.1371/journal.pcbi.1005629. eCollection 2017 Aug. PMID 28771616